CLINICAL TRIAL: NCT04561869
Title: Punctate Inner Choroidopathy (PIC) and Its Role in Progression of Pathological Myopia
Brief Title: PIC and Its Role in Progression of Pathological Myopia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shymaa kamel Ibrahim Hady, Assistant Lecture, Assiut University
Other Study IDs: PIC in Myopia
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-09

CONDITIONS: Punctate Inner Choroidopathy
MeSH Terms: conditions — White Dot Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Aim of the work PIC in pathological myopia has not been well documented due to difficult in diagnosis we conducted this retrospective study to characterize the clinical features of PIC in high myopic eye.

* To show the diagnostic criteria of PIC lesions in high myopic patients.
* Find out the prevalence of PIC related 'patchy atrophy'
* To determine risk factor for developed PIC in a series of highly myopic patients.
* Role of PIC in progression of high myopia.
* Calculate the progression rate of PIC related lesion, by the size change during follow-up.
* Search about complication of PIC in myopia. Patient and Methods This retrospective observational case series study included patients with high myopia who had been examined and followed-up in the High Myopia Clinic of the Tokyo Medical and Dental University. Approval from Ethics Committee of Tokyo Medical and Dental University was obtained, adhering to the tenets of Declaration of Helsinki. Signed informed consent documentation was obtained from all participants.

All study participants underwent a detailed ophthalmologic examination at baseline and at each follow-up visit. The examinations included measurements of best-corrected visual acuity (BCVA) using a Landolt C chart, refraction, slit lamp biomicroscopy, biometry for determination of axial length, (IOL Master; Carl Zeiss Meditec Co, Jena, Germany), fundus examination in medical mydriasis, fluorescein angiography, was performed with and colour fundus photography , and assessment of fundus autofluorescence (TRC-50DX; Topcon, Tokyo, Japan) a or the Heidelberg Spectralis HRA system. Swept source Optical coherence tomography (OCT) used in assessment of the RPE and photoreceptors using a (DRI-OCT;Topcon, Tokyo, Japan). As scanning protocols, 9 mm or 6 mm radial with 12 equal meridian scans were performed. The swept-source OCT device has an A-scan repetition rate of 100 000 Hz, and its light source operates in the wavelength range of 1 μm.

DETAILED DESCRIPTION:
Myopia The frequency of myopia and high myopia are growing on a worldwide for causes that not cleared. Myopia is vision challenges due to rises the risk of pathologic ophthalmic changes such as cataract, glaucoma, retinal detachment, and myopic macular degeneration, all of which can cause permanent vision loss.

High myopia was defined as an error of refractive above 8.0 diopters (D) or an axial length of 26.5 mm or more. Younger persons than 5 years, high myopia was defined by a refractive error of below- 4.0 D, and in children between 5 to 8 years, high myopia was defined by error of refraction below -6.0 D.

The term of pathologic myopia," "high myopia," and "axial myopia" have been used as a same in the literature. Pathologic myopia was defined as chorioretinal atrophy (by META-PM study group classification) with/or the existence of posterior staphylomas. Pathologic myopia is an significant origin of vision loss global, affecting up to 3% of the people. The effect of myopic maculopathy on impairment of vision is critical because the maculopathy is often affect both eye , permanent, and usually affects individuals in productive years.

Punctate inner choroidopathy Definition Punctate inner choroidopathy (PIC), classically bilateral and is considers one of "white dot syndromes" which usually presents with distinct ,multiple white-yellow lesions at posterior pole in the level of inner choroid and outer retina with a preference for young myopic female , without sign of old or recent anterior chamber or vitreous inflammation , with an increase the incidence of macular neovascularization (MNV).

ETIOLOGY The underlying pathophysiology are not completely understood. Multiple evanescent white dot syndrome( MEWDS)-like findings have been presented after traumatic subretinal bleeding, choroidal rupture, and penetrating injury or with angioid streaks, ensuring antigen exposure is likely causative factor. The present of acute retinopathy in Pseudoxanthoma elasticum (PXE) is marked along angioid streaks (breaks in the Bruch membrane), in which contact of retinal, RPE, and the Bruch membrane antigens to the immune system which stimulate an autoimmune system.

. Most inflammatory conditions in myopia are including the choriocapillaris. It can be suggested that weakness of the choriocapillaris due to anatomic changes in addition to unknown immunogenetic factors potentiate myopic eyes to primary inflammatory choriocapillaropathies.

CLINICAL FINDINGS Symptom Vision was usually slightly affected until the lesions were subfoveal or choroidal neovascular membranes developed.(8) According to the study by Gerstenblith and colleagues, initial symptoms in PIC are mostly scotoma (91%), blurred vision (86%), photopsia (73%), floaters (69%), photophobia (69%), and metamorphopsia (65%). Loss of peripheral vision was reported in 26% of patients. The consequence variable from return to the normal to bilateral profound loss of vision .

Sign Tools used in detecting and following PIC have involved fluorescein angiography, indocyanine green angiography, and OCT ,fundus autofluorescence (FAF) imaging and OCT angiography.

Fundoscopic features Small (100-300 microns), yellow-gray lesions (12-25 in number) which usually limited to the posterior pole and scattered in a haphazard (or rarely, linear) form.

The development of chorioretinal scars is frequency to occur as consequence at the sites of inflammation. Then, these scars become increasingly to well-defined ("punched out") and may come to be pigmented. These scars may progressively enlarge in size, leading to deterioration of symptoms over time.

OCT finding:

Stage I: minor irregularities change in the outer nuclear layer. Stage II: focal elevation of the retinal pigment epithelium/Bruch's membrane (RPE/BrM) complex with EZ and interdigitation zone disruption. Stage III: The lesion of moderate reflectivity breakdowns through the RPE and then grow to the dome of OPL through the photoreceptor layer. The RPE remain and BM at the break gradually disappear, exposing the choroidal part of the lesion. Stage IV: The lesion descends from the peak toward the choroidal part, subsequently a herniation of the OPL and inner retina (with a V-shaped change) through the defect in the RPE and BM. Stage V: The photoreceptor layer around the lesion is progressively missing with the drooping of the OPL and inner retina. This lead to V-shaped inward of the outer plexiform layer and inner retina into the choroid this is called "focal choroidal excavation .At the same time, RPE proliferation occurs (with posterior shadowing) to repair the RPE break so, the OPL framework reappear .

BM (Bruch's membrane); OPL (outer plexiform layer;) RPE ( retinal pigment epithelium), SD-OCT( spectral-domain optical coherence tomography).

fluorescein angiography (FA)& Indocyanine green angiography (ICG) FA in PIC patients show early hypofluorescence with late staining of inflammatory lesions, early hyperfluorescence can also happen, particularly if CNV is found. ICG shows midphase hypocyanescence at the posterior pole that may go beyond the lesions visible on FA and fundus.

Fundus autofluorescence (FAF) Active PIC lesions show hypoautofluorescent spots with a hyperautofluorescent border that disappear as the lesions regress. Atrophic PIC lesions display to be hypoautofluorescent.

Complication Serious visual loss occurs in about to 40% of patients mainly due to development of choroidal neovascularization (CNV). The Important associations of myopic choroidal neovascularization (MCNV) in highly myopic eyes with increasing levels of vascular endothelial growth factor or inflammatory cytokines and maculopathy lesions firmly indicate an association of inflammation in the cause of MCNVs.

Management The PIC management is tricky for multiple reasons. The varying in seriousness of disease between patients make that ideal l treatment range from observation to immunosuppression or intravitreal anti-VEGF therapy. The judgment whether a patient is benefit from maintenance therapy is hard due to the need to sense of balance between the varying outcome of patients with PIC and the hazards of immunosuppression. Large number of patients with PIC have prolonged times without disease activity and may go into long-standing remission, although in others these stable stages may be interrupted by unpredictable, sight-threatening episodes. Also, the evidence base to recommend any treatment approach is inadequate There is large difference between patients. So, mediation is necessary to treat new or active inflammatory "PIC" lesions especially when threatening the fovea, and to handle secondary CNV. Also, addition, the situation of the other eye requires attention.

The treatment options include local and systemic corticosteroids, systemic immunomodulatory drugs, intravitreal VEGF inhibitors (anti-VEGF), photodynamic therapy (PDT), argon laser, and submacular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Highly myopic patients.
* Men and women aged over 18 years
* Fundus changes typical of pathological myopia
* Minimum follow up period of 2 years

Exclusion Criteria:

* Another choroidal lesion other than MFC.
* Media opacity interfere with quality of image taking.
* Alternative diagnosis (especially other white dot syndromes or when it was unclear whether the lesions were due to pathologic myopia)
* If they had an underlying systemic condition that could mimic PIC (e.g., sarcoidosis, TB,)
* If they had history of travel to Histoplasma-endemic regions

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: we will enroll all high myopic patient with punctate inner choriodopathy lesion who have follow up period not less than 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic criteria of PIC in high or pathological myopic. | about 7 mounth
  Pick up the characteristic fundus feature and OCT finding of inflammatory lesion in pathological myopia cases
Calculate the progression rate of PIC related lesion. | about 7 mounth
  By measure the size of patchy atrophy changes during follow-up.
Development of complication as inflammatory choroidal neovascularization. | about 7 mounth
  Pick up the occurrence of inflammatory CNV during follow up period on fundus picture OCT images ,FA , and OCTA

SECONDARY OUTCOMES:
Prevalence of PIC in pathological myopia. | about 7 mounth
  The number of PIC patients in pathological myopia during this retrospective study of long follow up period
Final visual acuity. | about 7 mounth
  show the visual acuity of each patients at initial and last visits

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Kl Hady, As Lec, Principal Investigator — Department of Ophthalmology , Assiut University; Kyoko Oh Matsui, Prof, Study Chair — ,Department of Ophthalmology Tokyo Medical and Dental University; Omar Mo Ali, Prof, Study Chair — Department of Ophthalmology , Assiut University; Ehab Is Wasfi, As prof, Study Director — Department of Ophthalmology , Assiut University; Mahmoud Fa Rateb, As prof, Study Director — Department of Ophthalmology , Assiut University
Locations (1):
- Tokyo Medical and Dental University, Tokyo, Japan

REFERENCES:
- [Background] Flitcroft DI, He M, Jonas JB, Jong M, Naidoo K, Ohno-Matsui K, Rahi J, Resnikoff S, Vitale S, Yannuzzi L. IMI - Defining and Classifying Myopia: A Proposed Set of Standards for Clinical and Epidemiologic Studies. Invest Ophthalmol Vis Sci. 2019 Feb 28;60(3):M20-M30. doi: 10.1167/iovs.18-25957. PMID 30817826
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Fang Y, Yokoi T, Nagaoka N, Shinohara K, Onishi Y, Ishida T, Yoshida T, Xu X, Jonas JB, Ohno-Matsui K. Progression of Myopic Maculopathy during 18-Year Follow-up. Ophthalmology. 2018 Jun;125(6):863-877. doi: 10.1016/j.ophtha.2017.12.005. Epub 2018 Jan 19. PMID 29371011
- [Background] Niederer RL, Gilbert R, Lightman SL, Tomkins-Netzer O. Risk Factors for Developing Choroidal Neovascular Membrane and Visual Loss in Punctate Inner Choroidopathy. Ophthalmology. 2018 Feb;125(2):288-294. doi: 10.1016/j.ophtha.2017.09.002. Epub 2017 Oct 6. PMID 28993011
- [Background] Zarranz-Ventura J, Sim DA, Keane PA, Patel PJ, Westcott MC, Lee RW, Tufail A, Pavesio CE. Characterization of punctate inner choroidopathy using enhanced depth imaging optical coherence tomography. Ophthalmology. 2014 Sep;121(9):1790-7. doi: 10.1016/j.ophtha.2014.03.011. Epub 2014 May 20. PMID 24856311